CLINICAL TRIAL: NCT02045147
Title: Home Based Care Transitions Tailored by Cognition and Patient Activation: A Prudent Use of Transitional Care Resources
Brief Title: Home Based Care Transitions Tailored by Cognition and Patient Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0336-13-EP
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Disease
Keywords: Home Bound Care Transitions
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Grp 1a: Low Cognition, Low Activation (Experimental): Subjects will receive an 8 week care transition intervention with an Advanced Practice Registered Nurse-Nurse Practitioner (APRN-NP) and Certified Nursing Assistant (CNA). The APRN-NP will guide the care transition intervention. This group will receive the most intense intervention.
  Interventions: Behavioral: Grp 1a Low Cognition, Low Activation Intervention
- Grp 2a: Low Cognition, High Activation (Experimental): Subjects will receive an 8 week care transition intervention with an APRN-NP and CNA. The APRN-NP will guide the care transition intervention. This group will receive an intense intervention.
  Interventions: Behavioral: Grp 2a Low Cognition, High Activation Intervention
- Grp 3a: Normal Cognition, Low Activation (Experimental): Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  Interventions: Behavioral: Grp 3a Normal Cognition, Low Activation Intervention
- Grp 4a: Normal Cognition, High Activation (Experimental): Subjects will receive the least intensive intervention delivered by a RN coach.
  Interventions: Behavioral: Grp 4a Normal Cognition, High Activation Intervention
- Grp 1b: Low Cognition, Low Activation Usual Care (No Intervention): Comparison group to 1a intervention group
- Grp 2b Low Cognition, High Activation Usual Care (No Intervention): Comparison group to 2a intervention group
- Grp 3b: Normal Cognition, Low Activation Usual Care (No Intervention): Comparison group to 3a intervention group
- Grp 4b: Normal Cognition, High Activation Usual Care (No Intervention): Comparison group to 4a intervention group

INTERVENTIONS:
Behavioral: Grp 1a Low Cognition, Low Activation Intervention — The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation.
  Arms: Grp 1a: Low Cognition, Low Activation
Behavioral: Grp 2a Low Cognition, High Activation Intervention — The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation and handling stressful situations.
  Arms: Grp 2a: Low Cognition, High Activation
Behavioral: Grp 3a Normal Cognition, Low Activation Intervention — The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
  Arms: Grp 3a: Normal Cognition, Low Activation
Behavioral: Grp 4a Normal Cognition, High Activation Intervention — The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Focus is on maintaining behaviors during hardship and stress. Empowering, motivating and validating are strategies utilized.
  Arms: Grp 4a: Normal Cognition, High Activation

SUMMARY:
There is overwhelming evidence that patients with multiple chronic illnesses need better self-management skills. Discharge from the hospital may not be the most opportune time to be teaching patients these self-management skills. There are several different care transition models being used across the country; however we know that not every patient needs the same type or amount of an intervention. The purpose of this pilot study is to study the impact delivering a home based care transitions intervention (HBCTI) with four different groups tailored on cognition and level of patient activation compared to usual care (UC) resulting in 8 study arms on the outcomes of health care utilization (HCU) and health outcomes: patient-reported health status, assessment of care for chronic conditions, and health related quality of life in adult patients with multiple chronic diseases dismissed to home from an acute care facility. Our working hypothesis is that patients in the HBCTI groups compared to the UC groups will have lower HCU and improved outcomes (patient-reported health status, assessment of care for chronic conditions, and health related quality of life).

DETAILED DESCRIPTION:
One in five Medicare patients discharged from the hospital experience readmission within 30 days. Too often, hospital readmissions result from inadequate transition from hospital to home at discharge. Care transitions are complicated because of high patient acuity, multiple comorbidities, decreased length of stay, and multiple clinician involvement increasing the number of handoffs. With decreased length of stay, many patients do not comprehend or feel confident with instructions for discharge, thus management of their chronic illnesses are difficult. Most formal care transition programs are standardized and every patient receives similar strategies or interventions. However, it has been well documented that patients with cognitive problems and decreased activation are at high risk for re-hospitalization related to impaired self-management. We believe that assessment of cognition and patient activation during the patient's hospitalization will provide valuable information for discharge interventions. Data related to cognition and activation can be used to tailor discharge planning and help determine what type and how many resources are needed for individual patients after hospital discharge. The purpose of this feasibility study is to examine the impact of delivering a home based care transitions interventions (HBCTIs) with four different groups tailored on cognition and level of patient activation compared to usual care (UC) on the outcomes of health care utilization (HCU) and health outcomes: patient-reported health status, assessment of care for chronic conditions, and health related quality of life in adult patients with multiple chronic diseases discharged to home from the hospital.

We will test our intervention with the following aims: Aim 1.To evaluate the impact of HBCTIs on health care utilization. We will measure HCU (number of emergency department(ED) visits and number of readmissions) at 6 months after discharge. Our working hypothesis is that patients in the HBCTI groups compared to the UC groups will have lower HCU over time (6 months); Aim 2. To evaluate the impact of HBCTIs on the following health outcomes: patient-reported health status (PROMIS-29), assessment of care for chronic conditions (PACIC), and quality of life (EuroQol). Our working hypothesis is that patients in the HBCTI groups compared to the UC group will have improved patient-reported health status, assessment of care for chronic conditions, and quality of life (EuroQol) at 6 months after discharge.

The findings from this study have the potential to change this paradigm in three ways: 1) we will gain a better understanding of the role of cognition and patient activation in promoting self-management to enhance outcomes; 2). our innovative approach, which considers the unique needs of patients based on their level of cognition and patient activation will advance new concepts in care transition programs; 3) we will have a better understanding of varying intensities of visits, level of providers, and type and amount of strategies administered. This practical model for care transitions could serve as a model within the larger health care delivery system that could result in significant cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (age 19 and older) being discharged from the hospital with three or more chronic diseases;
* Have a score greater than 17 on the Montreal Cognitive Assessment (dementia);
* Reside within a 35 mile radius of Lincoln, Ne.; and
* Able to hear, speak and read English.

Exclusion Criteria:

Patients will be excluded if they:

* have a terminal illness;
* have a score of less than 17 on the Montreal Cognitive Assessment (dementia);
* are under the care of The Physicians Network (TPN) at St. Elizabeth Regional Medical Center (SERMC).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lani M Zimmerman, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Saint Elizabeth Regional Medical Center, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Grp 1a Low Cognition, Low Activation: Group 1: Subjects will receive an 8 week care transition intervention with an Advanced Practice Registered Nurse-Nurse Practitioner (APRN-NP) and Certified Nursing Assistant (CNA). The APRN-NP will guide the care transition intervention. This group will receive the most intense intervention.
  Grp 1 Low Cognition, Low Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation.
- Grp 2a Low Cognition, High Activation: Group 2: Subjects will receive an 8 week care transition intervention with an APRN-NP and CNA. The APRN-NP will guide the care transition intervention. This group will receive an intense intervention.
  Grp 2 Low Cognition, High Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation and handling stressful situations.
- Grp 3aNormal Cognition, Low Activation: Group 3: Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  Grp 3 Normal Cognition, Low Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
- Grp 4a Normal Cognition, High Activation: Group 4: Subjects will receive the least intensive intervention delivered by a RN coach.
  Grp 4 Normal Cognition, High Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Focus is on maintaining behaviors during hardship and stress. Empowering, motivating and validating are strategies utilized.
- Grp 1b Low Cognition, Low Activation: The comparison Group for Group 1a intervention group
- Grp 2b Low Cognition, High Activation: The comparison Group for Group 2a intervention group
- Grp 3b Normal Cognition, Low Activation: The comparison Group for Group 3a intervention group
- Grp 4b Normal Cognition, High Activation: The comparison group for Group 4a intervention group
Period: Overall Study
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3aNormal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation | Grp 2b Low Cognition, High Activation | Grp 3b Normal Cognition, Low Activation | Grp 4b Normal Cognition, High Activation
Started | 32 | 44 | 20 | 36 | 30 | 46 | 19 | 36
Completed | 21 | 32 | 20 | 34 | 27 | 36 | 19 | 33
Not Completed | 11 | 12 | 0 | 2 | 3 | 10 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Did not meet inclusion criteria at hospital discharge | 9 | 12 | 0 | 2 | 3 | 10 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis was completed on all patients that met inclusion criteria at discharge from the hospital.
Groups:
- Grp 1a Low Cognition, Low Activation: Subjects will receive an 8 week care transition intervention with an Advanced Practice Registered Nurse-Nurse Practitioner (APRN-NP) and Certified Nursing Assistant (CNA). The APRN-NP will guide the care transition intervention. This group will receive the most intense intervention.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation.
- Grp 2a Low Cognition, High Activation: Subjects will receive an 8 week care transition intervention with an APRN-NP and CNA. The APRN-NP will guide the care transition intervention. This group will receive an intense intervention.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation and handling stressful situations.
- Grp 3a Normal Cognition, Low Activation: Group 3a: Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
- Grp 4a Normal Cognition, High Activation: Subjects will receive the least intensive intervention delivered by a RN coach.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Focus is on maintaining behaviors during hardship and stress. Empowering, motivating and validating are strategies utilized.
- Grp 1b Low Cognition, Low Activation Usual Care: The comparison Group for Group 1a intervention group
- Grp 2b Low Cognition, High Activation Usual Care: The comparison Group for Group 2a intervention group
- Grp 4b Normal Cognition, High Activation Usual Care: The comparison group for Group 4a intervention group
- Total: Total of all reporting groups
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation | Grp 4b Normal Cognition, High Activation Usual Care | Total
Number analyzed (Participants) | 21 | 32 | 20 | 34 | 27 | 36 | 19 | 33 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 15 | 13 | 25 | 13 | 15 | 10 | 22 | 122
  >=65 years | 12 | 17 | 7 | 9 | 14 | 21 | 9 | 11 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (14.3) | 64.3 (13.8) | 55.9 (13.3) | 56.6 (14.7) | 66.1 (16.7) | 63.4 (16.1) | 59.3 (16.2) | 59.3 (13.3) | 61.3 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 10 | 25 | 10 | 18 | 13 | 17 | 131
  Male | 4 | 11 | 10 | 9 | 17 | 18 | 6 | 16 | 91
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 32 | 20 | 34 | 27 | 36 | 19 | 33 | 222

OUTCOME MEASURES:

1. Primary Outcome: Health Care Utilization
Description: Patient report of number of Emergency Department Visits and number of re-admissions to the hospital within a 6 month time period was measured. Validation data was obtained from the clinical sites.
Time Frame: 6 months
Population: Health care utilization was evaluated 6 months after intervention completion.
Measure: Number; unit: events
Groups:
- Grp 1a Low Cognition, Low Activation: Subjects will receive an 8 week care transition intervention with an Advanced Practice Registered Nurse-Nurse Practitioner (APRN-NP) and Certified Nursing Assistant (CNA). The APRN-NP will guide the care transition intervention. This group will receive the most intense intervention.
  Grp 1 Low Cognition, Low Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation.
- Grp 2a: Low Cognition, High Activation: Subjects will receive an 8 week care transition intervention with an APRN-NP and CNA. The APRN-NP will guide the care transition intervention. This group will receive an intense intervention.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation and handling stressful situations.
- Grp 3a: Normal Cognition, Low Activation: Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
- Grp 4a; Normal Cognition, High Activation: Group 4: Subjects will receive the least intensive intervention delivered by a RN coach.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Focus is on maintaining behaviors during hardship and stress. Empowering, motivating and validating are strategies utilized.
- Grp 1b: Low Cognition, Low Activation Usual Care: The comparison Group for Group 1a intervention group
- Grp 2b: Low Cognition, High Activation Usual Care: The comparison Group for Group 2a intervention group
- Grp 3b: Normal Cognition, Low Activation Usual Care: The comparison Group for Group 3a intervention group
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a: Low Cognition, High Activation | Grp 3a: Normal Cognition, Low Activation | Grp 4a; Normal Cognition, High Activation | Grp 1b: Low Cognition, Low Activation Usual Care | Grp 2b: Low Cognition, High Activation Usual Care | Grp 3b: Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 21 | 32 | 20 | 34 | 27 | 36 | 19 | 33
events
  Emergency Department visits | 7 | 8 | 4 | 3 | 5 | 13 | 8 | 10
  Readmissions | 5 | 7 | 8 | 6 | 4 | 11 | 5 | 11

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Pain Interference
Description: Pain interference is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Assessing patient perception of pain interference is measured as a 4-item short form scale on the PROMIS-29 survey. Each item is scored from 1-5 with a 1 indicating "not at all" and 5 indicating "very much." The T-Score for the average general population is 50. Higher scores mean more pain interference, thus a worse outcome. A score change of 2-3 points has been reported as clinically meaningful differences.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Grp 4a: Normal Cognition, High Activation: Subjects will receive the least intensive intervention delivered by a RN coach.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Focus is on maintaining behaviors during hardship and stress. Empowering, motivating and validating are strategies utilized.
- Grp 3b Normal Cognition, Low Activation Usual Care: The comparison Group for Group 3a intervention group
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a: Low Cognition, High Activation | Grp 3a: Normal Cognition, Low Activation | Grp 4a: Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 20 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 58.8 (9.8) | 57.0 (11.5) | 61.4 (10.9) | 54.2 (8.5) | 56.0 (11.0) | 55.4 (11.0) | 56.6 (10.9) | 52.4 (9.2)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.463, t-test, 2 sided; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-4.98 to 10.65], Standard Error of Mean 3.82
Statistical Analysis 2: Comparison: Grp 2a: Low Cognition, High Activation vs Grp 2b Low Cognition, High Activation Usual Care; Test type: Other; p = 0.634, t-test, 2 sided; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-5.23 to 8.49], Standard Error of Mean 3.40
Statistical Analysis 3: Comparison: Grp 3a: Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.259, t-test, 2 sided; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-3.74 to 13.32], Standard Error of Mean 4.15
Statistical Analysis 4: Comparison: Grp 4a: Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.472, t-test, 2 sided; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-3.21 to 6.84], Standard Error of Mean 2.50

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System-Physical Functioning
Description: Physical Functioning is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Physical functioning is measured as a 4-item short form subscale on the PROMIS-29 survey. The patients' answers to the Physical Functioning items are scored from 1-5, with a 1 indicating "unable to do" and 5 indicating "without any difficulty." Each subscales forms its own score subscale measures are scored on the T-score metric. High scores indicating better or higher physical functioning
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Grp 1a: Low Cognition, Low Activation: Subjects will receive an 8 week care transition intervention with an Advanced Practice Registered Nurse-Nurse Practitioner (APRN-NP) and Certified Nursing Assistant (CNA). The APRN-NP will guide the care transition intervention. This group will receive the most intense intervention.
  Grp 1 Low Cognition, Low Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided at a 5th grade reading level. The "teach back" method is used to validate knowledge, skills and confidence. Once knowledge is validated, the interventions focused on motivation.
- Grp 3a Normal Cognition, Low Activation: Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
Arm/Group | Grp 1a: Low Cognition, Low Activation | Grp 2a: Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a: Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b: Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 39.1 (9.2) | 42.1 (10.2) | 36.3 (10.4) | 43.6 (8.6) | 41.1 (8.1) | 43.8 (9.2) | 40.8 (9.4) | 44.5 (10.6)
Statistical Analysis 1: Comparison: Grp 1a: Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.532, t-test, 2 sided; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-8.5 to 4.5], Standard Error of Mean 3.15
Statistical Analysis 2: Comparison: Grp 2a: Low Cognition, High Activation vs Grp 2b: Low Cognition, High Activation Usual Care; Test type: Other; p = 0.574, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-7.5 to 4.2], Standard Error of Mean 2.9
Statistical Analysis 3: Comparison: Grp 3a Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.254, t-test, 2 sided; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-12.3 to 3.4], Standard Error of Mean 3.8
Statistical Analysis 4: Comparison: Grp 4a: Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.759, t-test, 2 sided; Mean Difference (Final Values) = -.9, 95% CI 2-sided [-6.3 to 4.6], Standard Error of Mean 2.7

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System-Satisfaction With Social Roles
Description: Ability to participate in social roles and activities is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Ability to participate in social roles and activities is measured as a 4-item short form subscale on the PROMIS-29 survey. The patients' answers to the PROMIS-29 are scored from 1-5, with a 1 indicating "never" and 5 indicating "always." Each subscales forms its own score subscale measures are scored on the T-score metric. High scores indicating more ability to participate in social roles and activities.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Grp 3a; Normal Cognition, Low Activation: Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
Arm/Group | Grp 1a: Low Cognition, Low Activation | Grp 2a: Low Cognition, High Activation | Grp 3a; Normal Cognition, Low Activation | Grp 4a: Normal Cognition, High Activation | Grp 1b: Low Cognition, Low Activation Usual Care | Grp 2b: Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 19 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 49.3 (11.3) | 49.2 (10.7) | 43.8 (10.5) | 50.4 (11.1) | 44.1 (8.4) | 50.4 (10.9) | 43.3 (6.5) | 52.8 (11.1)
Statistical Analysis 1: Comparison: Grp 1a: Low Cognition, Low Activation vs Grp 1b: Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.153, t-test, 2 sided; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-2.1 to 12.7], Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Grp 2a: Low Cognition, High Activation vs Grp 2b: Low Cognition, High Activation Usual Care; Test type: Other; p = 0.729, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-7.9 to 5.5], Standard Error of Mean 3.3
Statistical Analysis 3: Comparison: Grp 3a; Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.886, t-test, 2 sided; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-6.6 to 7.6], Standard Error of Mean 3.5
Statistical Analysis 4: Comparison: Grp 4a: Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.446, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-8.7 to 3.9], Standard Error of Mean 3.1

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System- Anxiety
Description: Anxiety is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Assessing patient anxiety is measured as a 4-item short form subscale on the PROMIS-29 survey. The patients' answers to the PROMIS-29 are scored from 1-5, with a 1 indicating "never" and 5 indicating "always." Each subscales forms its own score subscale measures are scored on the T-score metric. High scores indicating more anxiety and a worse outcome, and lower scores are indicative of less anxiety and a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Grp 1a: Low Cognition, Low Activation | Grp 2a: Low Cognition, High Activation | Grp 3a: Normal Cognition, Low Activation | Grp 4a: Normal Cognition, High Activation | Grp 1b: Low Cognition, Low Activation Usual Care | Grp 2b: Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 54.0 (12.7) | 51.0 (7.8) | 53.5 (11.7) | 46.6 (9.1) | 51.3 (9.8) | 46.8 (10.1) | 53.1 (10.7) | 48.1 (7.7)
Statistical Analysis 1: Comparison: Grp 1a: Low Cognition, Low Activation vs Grp 1b: Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.521, t-test, 2 sided; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-5.7 to 11.1], Standard Error of Mean 4.1
Statistical Analysis 2: Comparison: Grp 2a: Low Cognition, High Activation vs Grp 2b: Low Cognition, High Activation Usual Care; Test type: Other; p = 0.146, t-test, 2 sided; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-1.5 to 9.5], Standard Error of Mean 2.7
Statistical Analysis 3: Comparison: Grp 3a: Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.926, t-test, 2 sided; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-8.5 to 9.3], Standard Error of Mean 4.3
Statistical Analysis 4: Comparison: Grp 4a: Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.526, t-test, 2 sided; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-6.4 to 3.3], Standard Error of Mean 2.4

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System-Fatigue
Description: Fatigue is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Fatigue is measured as a 4-item short form subscale on the PROMIS-29 survey. The patients' answers to the PROMIS-29 are scored from 1-5, with a 1 indicating "not at all" and 5 indicating "very much." Each subscales forms its own score subscale measures are scored on the T-score metric. High scores indicating more fatigue and a worse outcome and lower scores are indicative of less fatigue and a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Grp 4 Normal Cognition, High Activation: Group 4: Subjects will receive the least intensive intervention delivered by a RN coach.
  Grp 4 Normal Cognition, High Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Focus is on maintaining behaviors during hardship and stress. Empowering, motivating and validating are strategies utilized.
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4 Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 54.8 (10.9) | 54.3 (11.0) | 56.7 (12.2) | 50.5 (10.5) | 55.9 (10.5) | 49.3 (11.2) | 59.1 (8.5) | 48.0 (8.3)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.776, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-9.2 to 6.9], Standard Error of Mean 3.9
Statistical Analysis 2: Comparison: Grp 2a Low Cognition, High Activation vs Grp 2b Low Cognition, High Activation Usual Care; Test type: Other; p = 0.135, t-test, 2 sided; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [-1.6 to 11.7], Standard Error of Mean 3.3
Statistical Analysis 3: Comparison: Grp 3a Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.556, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-10.9 to 6.0], Standard Error of Mean 4.1
Statistical Analysis 4: Comparison: Grp 4 Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.361, t-test, 2 sided; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-2.9 to 7.9], Standard Error of Mean 2.7

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System- Depression
Description: Depression is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Depression is measured as a 4-item short form subscale on the PROMIS-29 survey. The patients' answers to the PROMIS-29 are scored from 1-5, with a 1 indicating "never" and 5 indicating "always." Each subscales forms its own score subscale measures are scored on the T-score metric. High scores indicating more feeling of depression and a worse outcome and lower scores are indicative of less depression and a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 55.2 (10.9) | 50.5 (10.4) | 54.4 (11.0) | 49.4 (9.1) | 52.6 (12.9) | 47.4 (10.1) | 53.3 (8.2) | 48.7 (8.0)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.564, t-test, 2 sided; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-6.4 to 11.6], Standard Error of Mean 4.4
Statistical Analysis 2: Comparison: Grp 2a Low Cognition, High Activation vs Grp 2b Low Cognition, High Activation Usual Care; Test type: Other; p = 0.307, t-test, 2 sided; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-3.0 to 9.3], Standard Error of Mean 3.1
Statistical Analysis 3: Comparison: Grp 3a Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.768, t-test, 2 sided; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-6.7 to 8.9], Standard Error of Mean 3.8
Statistical Analysis 4: Comparison: Grp 4a Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.785, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-4.2 to 5.5], Standard Error of Mean 2.4

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System-Sleep Deprivation
Description: Sleep disturbance is one of the 7 domains of the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS-29 is the shortest profile, with 4 questions asked for each of 7 domains, plus the single pain intensity item. PROMIS measures are scored on the T-score metric. Each short form is scored separately, yielding a total of 7 domain scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. There is no total score, but each axis forms its own score.
  Assessing sleep disturbance is measured as a 4-item short form subscale on the PROMIS-29 survey. The patients' answers to the sleep disturbance domain are scored from 1-5, with a 1 indicating "very good or very much" and 5 indicating "very poor or not at all." High scores indicating more sleep disturbance and a worse outcome, and lower scores are indicative of less sleep disturbance and a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Grp 4b High Cognition, High Activation Usual Care: The comparison Group for Group 4a intervention group
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b High Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 50.1 (9.3) | 51.5 (10.7) | 53.5 (9.1) | 48.4 (10.3) | 50.5 (9.6) | 46.9 (11.7) | 52.4 (9.7) | 46.6 (9.2)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.917, t-test, 2 sided; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-7.5 to 6.8], Standard Error of Mean 3.5
Statistical Analysis 2: Comparison: Grp 2a Low Cognition, High Activation vs Grp 2b Low Cognition, High Activation Usual Care; Test type: Other; p = 0.181, t-test, 2 sided; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-2.2 to 11.3], Standard Error of Mean 3.3
Statistical Analysis 3: Comparison: Grp 3a Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.772, t-test, 2 sided; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-6.3 to 8.3], Standard Error of Mean 3.6
Statistical Analysis 4: Comparison: Grp 4a Normal Cognition, High Activation vs Grp 4b High Cognition, High Activation Usual Care; Test type: Other; p = 0.526, t-test, 2 sided; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-3.8 to 7.3], Standard Error of Mean 2.8

9. Secondary Outcome: Patient Assessment of Chronic Illness Care
Description: The Patient Assessment of Chronic Illness Care (PACIC) Survey is a 20-item patient report instrument that assesses patient's receipt of clinical services and actions consistent with the Chronic Care Model. Respondents rate how often they experienced the content described in the item on a 5-point scale ranging from 1 (no or never) to 5 (yes or always). Patients rated the care received from their health care team. The PACIC consists of 5 scales and an overall summary score, each having good internal consistency for brief scales. The five subscales were Patient Activation; Delivery System/ Decision Support; Goal Setting; Problem-solving/Contextual Counseling; and Follow-up/ Coordination. Overall mean summary score (range 1-5) was used in analysis. Higher scores are more positive rating of their receipt of clinical services.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 20 | 16 | 25 | 16 | 22 | 12 | 20
score on a scale | 2.9 (1.2) | 2.9 (1.0) | 2.5 (1.0) | 3.0 (1.0) | 2.8 (1.1) | 3.2 (.9) | 2.5 (1.0) | 2.6 (.9)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.872, t-test, 2 sided; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.8 to .9], Standard Error of Mean .42
Statistical Analysis 2: Comparison: Grp 2a Low Cognition, High Activation vs Grp 2b Low Cognition, High Activation Usual Care; Test type: Other; p = 0.387, t-test, 2 sided; Mean Difference (Final Values) = -.3, 95% CI 2-sided [-.87 to .34], Standard Error of Mean .30
Statistical Analysis 3: Comparison: Grp 3a Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.916, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-.37 to .81], Standard Error of Mean .38
Statistical Analysis 4: Comparison: Grp 4a Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.189, t-test, 2 sided; Mean Difference (Final Values) = .4, 95% CI 2-sided [-.19 to .94], Standard Error of Mean .28

10. Secondary Outcome: Health Related Quality of Life EuroQol-5D (EQ-5D)
Description: Quality of life was measured by the EuroQol-5 (EQ-5D) and consists of 1 question for each of the 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Patients indicate their health state for each of the 5 dimensions. The 5 responses give a health state represented by a 5-digit number (for example, 12231) corresponding to response categories reported by patients for the dimensions. Health states are scored to give the EQ-5D-5L index using a scoring algorithm from a value set derived from valuation tasks typically undertaken with general population samples. The five dimensions are combined into a 5-digit number that describes the patient's health state. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation Usual Care | Grp 2b Low Cognition, High Activation Usual Care | Grp 3b Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 13 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 0.68 (0.24) | 0.76 (0.14) | 0.65 (0.17) | 0.80 (0.09) | 0.72 (0.20) | 0.77 (0.19) | 0.76 (0.08) | 0.80 (0.11)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b Low Cognition, Low Activation Usual Care; Test type: Other; p = 0.627, t-test, 2 sided; Mean Difference (Final Values) = -.04, 95% CI 2-sided [-.21 to .13], Standard Error of Mean .08
Statistical Analysis 2: Comparison: Grp 2a Low Cognition, High Activation vs Grp 2b Low Cognition, High Activation Usual Care; Test type: Other; p = 0.840, t-test, 2 sided; Mean Difference (Final Values) = -.01, 95% CI 2-sided [-.11 to .09], Standard Error of Mean .05
Statistical Analysis 3: Comparison: Grp 3a Normal Cognition, Low Activation vs Grp 3b Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.049, t-test, 2 sided; Mean Difference (Final Values) = -.11, 95% CI 2-sided [-.22 to -.00], Standard Error of Mean .05
Statistical Analysis 4: Comparison: Grp 4a Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.952, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-.06 to .06], Standard Error of Mean .03

11. Secondary Outcome: EQ-5D Visual Analog Scale (VAS)
Description: Used alongside the EuroQol-5D (EQ-5D), the EQ visual analog scale (VAS) is a 20 cm VAS "assessing your own health today" with endpoints labeled "Best imaginable health state" (100) and "Worst imaginable health state" (0). EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a: Low Cognition, High Activation | Grp 3a: Normal Cognition, Low Activation | Grp 4a; Normal Cognition, High Activation | Grp 1b: Low Cognition, Low Activation Usual Care | Grp 2b: Low Cognition, High Activation Usual Care | Grp 3b: Normal Cognition, Low Activation Usual Care | Grp 4b Normal Cognition, High Activation Usual Care
Number analyzed (Participants) | 14 | 21 | 16 | 26 | 16 | 24 | 12 | 24
score on a scale | 68.2 (28.3) | 67.2 (27.2) | 62.4 (23.0) | 73.5 (18.3) | 61.3 (19.6) | 79.0 (17.3) | 72.9 (13.4) | 77.2 (13.0)
Statistical Analysis 1: Comparison: Grp 1a Low Cognition, Low Activation vs Grp 1b: Low Cognition, Low Activation Usual Care; Test type: Other; p = .436, t-test, 2 sided; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [-11.07 to 25.00]
Statistical Analysis 2: Comparison: Grp 2a: Low Cognition, High Activation vs Grp 2b: Low Cognition, High Activation Usual Care; Test type: Other; p = .088, t-test, 2 sided; Mean Difference (Final Values) = -11.8, 95% CI 2-sided [-25.24 to 1.80], Standard Error of Mean 6.71
Statistical Analysis 3: Comparison: Grp 3a: Normal Cognition, Low Activation vs Grp 3b: Normal Cognition, Low Activation Usual Care; Test type: Other; p = 0.169, t-test, 2 sided; Median Difference (Final Values) = -10.5, 95% CI 2-sided [-25.86 to 4.77], Standard Error of Mean 7.45
Statistical Analysis 4: Comparison: Grp 4a; Normal Cognition, High Activation vs Grp 4b Normal Cognition, High Activation Usual Care; Test type: Other; p = 0.416, t-test, 2 sided; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-12.79 to 5.37], Standard Error of Mean 4.52

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Grp 3a Normal Cognition, Low Activation: Group 3: Subjects will receive an 4 week care transition intervention with a Registered Nurse (RN) Coach. This group will be evaluated at four weeks, if the patient activation levels are still low, they will be referred to the 4 week APRN-NP and CNA.
  Grp 3 Normal Cognition, Low Activation: The intervention is focused on knowledge, skills, confidence and creating a partnership with the health care provider. Education is provided for areas of misunderstanding. The "teach back" method is used to validate knowledge, skills and confidence. Interventions are focused on motivation and developing personal behavioral goals.
Arm/Group | Grp 1a Low Cognition, Low Activation | Grp 2a Low Cognition, High Activation | Grp 3a Normal Cognition, Low Activation | Grp 4a Normal Cognition, High Activation | Grp 1b Low Cognition, Low Activation | Grp 2b Low Cognition, High Activation | Grp 3b Normal Cognition, Low Activation | Grp 4b Normal Cognition, High Activation
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/32 | 0/20 | 0/34 | 0/27 | 0/36 | 0/19 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/32 | 0/20 | 0/34 | 0/27 | 0/36 | 0/19 | 0/33
Other Adverse Events (participants affected / at risk) | 0/21 | 0/32 | 0/20 | 0/34 | 0/27 | 0/36 | 0/19 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes